CLINICAL TRIAL: NCT00522236
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, Adjuvanted Influenza Vaccine, Formulation 2007-2008, When Administered to Elderly Subjects
Brief Title: Safety and Immunogenicity of a Commercially Available Influenza Vaccine (Formulation 2007/2008) When Administered to Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70P5S; 2007-000966-19
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: Adjuvanted Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Antigens, Surface

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: Surface Antigen, Inactivated, Adjuvanted Influenza Vaccine, Formulation 2007-2008

INTERVENTIONS:
Biological: Surface Antigen, Inactivated, Adjuvanted Influenza Vaccine, Formulation 2007-2008 — A single 0.5mL dose of Novartis adjuvanted subunit influenza vaccine, Fluad contained 45μg of viral hemagglutinin, composed of 15μg of the three influenza antigens:
  * A(H1N1) strain: IVR-145 (Solomon Island/3/2006 - like strain)
  * A(H3N2) strain: NYMC X-161B (A/Wisconsin/67/2005-like strain)
  * B strain: (B/Malaysia/2506/2004-like strain) in accordance with the recommendations of the World Health Organization, the EU and the national Regulatory Agencies for the 2007/2008 season.
  The vaccine is a milky liquid, and was packaged in ready to use, single dose syringes.
  A single dose of FLUAD vaccine was administered intramuscularly, preferably in the deltoid muscle of the non dominant arm.

SUMMARY:
To evaluate the antibody response to each influenza vaccine antigen when administering a single dose to subjects aged 65 years and over

ELIGIBILITY:
Inclusion Criteria:

- 65 years of age or older

Exclusion Criteria:

* any serious disease such as cancer, autoimmune disease, advanced arteriosclerotic disease or insulin-dependent diabetes mellitus, chronic obstructive pulmonary disease (COPD) that requires oxygen therapy, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure and bleeding diathesis or conditions associated with prolonged bleeding time
* hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or kanamycin or any other component of the vaccine
* history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
* known or suspected (or high risk of developing) impairment/alteration of immune function
* any acute disease or infections requiring systemic antibiotic or antiviral therapy within the past 7 days
* fever within the past 3 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Antibody response to each influenza vaccine antigen as measured by Single Radial Hemolysis in elderly subjects (≥65y) in compliance with the requirements of the current EU recommendations for a new formulation of a licensed flu vaccine (CPMP/BWP/214/96) | 21 days post-vaccination
  The measures of immunogenicity for each antigen are:
  * the geometric mean area (GMA) on Day 0 and Day 21
  * the Day 21/Day 0 geometric mean area ratio (GMR)
  * the percentage of subjects achieving seroconversion1 or significant increase in antibody titer2
  * the percentage of subjects achieving an SRH area ≥ 25 mm2 on Day 0 and Day 21
    1. Seroconversion is defined as negative prevaccination serum/postvaccination serum area ≥ 25 mm2.
    2. Significant increase in antibody titer is defined as at least a 50% increase in area.

SECONDARY OUTCOMES:
To evaluate the safety of the administration of a single intramuscular (IM) injection of FLUAD® vaccine (formulation 2007/2008) in elderly subjects (≥ 65 years). | 3 days, respectively 21 days post-vaccination
  Number and percentage of subjects with at least one local reaction between Day 0 and Day 3 after vaccine injection.
  Number and percentage of subjects with at least one systemic reaction between Day 0 and Day 3 after vaccine injection.
  Number and percentage of subjects with at least one adverse event between Day 0 and the study termination visit (Day 21, window: 20-24).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (2):
- Italy (2):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Chieti
  - Ufficio Igiene e Sanità Pubblica di Lanciano, ASL Lanciano - Vasto, Via S. Spaventa, 37, Lanciano